CLINICAL TRIAL: NCT01528514
Title: The Effects of CUrcuminoids on Coronary Artery byPass graftIng-related myocarDial Infarction Study
Brief Title: Effects of CUrcuminoids on Coronary Artery byPass graftIng-related myocarDial Infarction Study
Acronym: CUPID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wanwarang Wongcharoen, MD. (Other)
Responsible Party: Sponsor-Investigator, Wanwarang Wongcharoen, MD., Principal investigator, Thailand Research Fund
Organization: Thailand Research Fund (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRG5380258
Record Dates: First submitted 2012-01-31; First posted 2012-02-08 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Coronary Artery Bypass Grafting
Keywords: Myocardial infarction; Coronary artery bypass grafting; Anti-oxidant; Curcuminoids
MeSH Terms: conditions — Myocardial Infarction | interventions — Diarylheptanoids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Curcuminoids (Active Comparator)
  Interventions: Dietary Supplement: Curcuminoids
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Curcuminoids — Curcuminoids in capsule form, 4 capsules four times daily (4 grams/day)
  Arms: Curcuminoids
Other: Placebo — Placebo in capsule form, 4 capsules 4 times/day
  Arms: Placebo

SUMMARY:
It is well-established that myocardial infarction (MI) associated with coronary artery bypass graft surgery (CABG) predicts the poor outcome. Nevertheless, the cardioprotective therapies to limit myocardial injury after CABG are lacking. Previous studies have shown that curcuminoids suppress pro-inflammatory cytokines during cardiopulmonary bypass surgery and decrease the occurrence of cardiomyocytic apoptosis after cardiac ischemia/reperfusion injury in animal models. The investigators aim to evaluate whether curcuminoids prevent MI after CABG, compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing CABG without valve surgery

Exclusion Criteria:

* emergency cardiac surgery
* any increase in CK-MB above upper limit of normal range (ULN) at the time of randomization
* patients with cholestatic jaundice (total bilirubin > 2-fold ULN)
* severe liver disease (AST or ALT > 3-fold ULN)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative myocardial infarction | participants will be followed for the duration of hospital stay, an expected average of 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Wanwarang Wongcharoen, MD, Principal Investigator — Faculty of Medicine, Chiang Mai University
Locations (1):
- Maharaj Nakorn Chiang Mai hospital, Chiang Mai, Thailand